CLINICAL TRIAL: NCT00000555
Title: Women's Angiographic Vitamin and Estrogen Trial (WAVE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 99; N01HV68165 (NIH); N01HV68166 (NIH); N01HV68167 (NIH); N01HV68168 (NIH); N01HV68169 (NIH); N01HV68170 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2005-08

CONDITIONS: Cardiovascular Diseases; Coronary Arteriosclerosis; Coronary Disease; Heart Diseases; Myocardial Ischemia; Postmenopause
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — Estrogen Replacement Therapy; Estrogens, Conjugated (USP); Progesterone; Hormone Replacement Therapy; Dietary Supplements; Food; Ascorbic Acid; Vitamin E

INTERVENTIONS:
Drug: estrogen replacement therapy
Drug: estrogens, conjugated
Drug: progesterone
Drug: hormone replacement therapy
Drug: supplementation, food
Drug: ascorbic acid
Drug: vitamin e

SUMMARY:
To assess whether hormonal replacement therapy and/or antioxidant treatment would stabilize or inhibit progression, and induce regression of coronary plaques. The mechanisms by which these treatments modified atherosclerosis in women were also explored.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary artery disease is the leading cause of death in the United States, accounting for over 500,000 deaths each year. Although the onset of coronary artery disease is delayed in women, it is the single most important cause of death in women over the entire life span. Indeed, because more women than men survive to old age, mortality due to coronary artery disease for all ages combined is as great in women as in men. Furthermore, once they present with clinical evidence of coronary artery disease, women have a prognosis as poor as, or even worse, than that for men. In part, this may be due to late recognition of coronary artery disease in women, less intensive treatment of women, or a more adverse risk profile in women who develop coronary artery disease. The report of a recent Working Group on Angiographic Trials of Atherosclerosis Prevention notes that, compared to males, females who develop coronary artery disease, have various different characteristics which may affect the vascular response to lipid-altering interventions. These differences led the report to question whether the mechanisms and clinical benefits of lipid-altering agents may be different in men and women. It further noted that angiographic trials conducted to date have been based primarily upon the cholesterol-lowering treatments of diet or drugs and suggested that other approaches based upon the lipid hypothesis could profitably be tested and should be given the highest priority at this time; specifically recommended were trials of hormone replacement and antioxidant therapy in women.

DESIGN NARRATIVE:

Subjects were randomized into a 2 x 2 factorial trial of hormone replacement therapy and antioxidant therapy. Women were randomized into four treatment groups: both active hormone replacement and antioxidant; active hormone replacement therapy and antioxidant placebo; active antioxidant therapy and hormone replacement placebo; double placebo plus usual care. Hormone replacement therapy consisted of estrogen plus a progestin (PremPro) for all gynecologically intact women, and unopposed estrogen (Premarin) for women with hysterectomies. Antioxidants consisted of a combination of vitamin E and vitamin C. Angiographic change was a primary endpoint of this trial. The study was double-blind to the extent permitted by the interventions; however, it was fully-blinded with respect to outcome variables. Recruitment ended in August 1999. The mean duration of follow-up was approximately three years.

The NHLBI awarded R01HL68397 in April 2001 as an ancillary study to WAVE. The study entitled "Modifying Oxidative Damage in WAVE" has its on site on this database.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Postmenopausal women, up to age 86, with angiographically documented coronary artery disease of at least 15 percent, but no more than 75 percent occlusion.

Ages: 38 Years to 86 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-08; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Verter — George Washington University

REFERENCES:
- [Background] Waters DD, Alderman EL, Hsia J, Howard BV, Cobb FR, Rogers WJ, Ouyang P, Thompson P, Tardif JC, Higginson L, Bittner V, Steffes M, Gordon DJ, Proschan M, Younes N, Verter JI. Effects of hormone replacement therapy and antioxidant vitamin supplements on coronary atherosclerosis in postmenopausal women: a randomized controlled trial. JAMA. 2002 Nov 20;288(19):2432-40. doi: 10.1001/jama.288.19.2432. PMID 12435256
- [Background] Hsia J, Alderman EL, Verter JI, Rogers WJ, Thompson P, Howard BV, Cobb FR, Ouyang P, Tardif JC, Higginson L, Bittner V, Barofsky I, Steffes M, Gordon DJ, Proschan M, Younes N, Waters D. Women's angiographic vitamin and estrogen trial: design and methods. Control Clin Trials. 2002 Dec;23(6):708-27. doi: 10.1016/s0197-2456(02)00237-4. PMID 12505248
- [Background] Hsia J, Bittner V, Tripputi M, Howard BV. Metabolic syndrome and coronary angiographic disease progression: the Women's Angiographic Vitamin & Estrogen trial. Am Heart J. 2003 Sep;146(3):439-45. doi: 10.1016/S0002-8703(03)00227-8. PMID 12947360
- [Background] Howard BV, Hsia J, Ouyang P, Van Voorhees L, Lindsay J, Silverman A, Alderman EL, Tripputi M, Waters DD. Postmenopausal hormone therapy is associated with atherosclerosis progression in women with abnormal glucose tolerance. Circulation. 2004 Jul 13;110(2):201-6. doi: 10.1161/01.CIR.0000134955.93951.D5. Epub 2004 Jun 28. PMID 15226212
- [Background] Levy AP, Friedenberg P, Lotan R, Ouyang P, Tripputi M, Higginson L, Cobb FR, Tardif JC, Bittner V, Howard BV. The effect of vitamin therapy on the progression of coronary artery atherosclerosis varies by haptoglobin type in postmenopausal women. Diabetes Care. 2004 Apr;27(4):925-30. doi: 10.2337/diacare.27.4.925. PMID 15047650
- [Background] Bittner V, Tripputi M, Hsia J, Gupta H, Steffes M; Women's Angiographic Vitamin & Estrogen Investigators. Remnant-like lipoproteins, hormone therapy, and angiographic and clinical outcomes: the Women's Angiographic Vitamin & Estrogen Trial. Am Heart J. 2004 Aug;148(2):293-9. doi: 10.1016/j.ahj.2004.01.025. PMID 15308999
- [Background] Kelemen M, Vaidya D, Waters DD, Howard BV, Cobb F, Younes N, Tripputti M, Ouyang P. Hormone therapy and antioxidant vitamins do not improve endothelial vasodilator function in postmenopausal women with established coronary artery disease: a substudy of the Women's Angiographic Vitamin and Estrogen (WAVE) trial. Atherosclerosis. 2005 Mar;179(1):193-200. doi: 10.1016/j.atherosclerosis.2004.09.021. Epub 2004 Dec 28. PMID 15721027
- [Background] Ruo B, Tripputi MT, Hsue PY, Saigo M, Ouyang P, Waters DD. Usefulness of serum endothelin levels in predicting death and myocardial infarction but not coronary progression in postmenopausal women with coronary disease (from the Women's Angiographic Vitamin and Estrogen [WAVE] study). Am J Cardiol. 2005 Aug 1;96(3):335-8. doi: 10.1016/j.amjcard.2005.03.071. PMID 16054453
- Available data/document: Individual Participant Data Set: WAVE — http://biolincc.nhlbi.nih.gov/studies/wave/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/wave/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/wave/
- Available data/document: Manual of Procedures — http://biolincc.nhlbi.nih.gov/studies/wave/